CLINICAL TRIAL: NCT00463034
Title: Genetic Factors Affecting Breast Cancer Progression
Brief Title: Genes That Affect Disease Progression in Women With Newly Diagnosed or Metastatic Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sheffield (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000540737; SHEFF-05/Q2308/15; SHEFF-USMS-05/Q2308/15; EU-20726; SHEFF-STH13824; SHEFF-106364; GENFABRCA
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2008-11

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Microarray Analysis; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis; Chromatography, High Pressure Liquid; Immunohistochemistry

INTERVENTIONS:
Genetic: microarray analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: high performance liquid chromatography
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and help doctors understand how patients respond to treatment.

PURPOSE: This clinical trial is assessing how changes in genes affect disease progression in women with newly diagnosed or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Correlate inherited and acquired variations in candidate genes with breast cancer progression and survival in women with newly diagnosed or metastatic breast cancer.

Secondary

* Establish a repository of blood and tumor samples from these patients, linked to a database of clinical, pathological, and treatment outcome data for future research studies.

OUTLINE: Patients complete epidemiological questionnaires and undergo blood sample collection. Tumor tissue specimens are requested from the pathology departments.

Blood samples are analyzed for single nucleotide polymorphisms and other polymorphic variants in candidate genes by polymerase chain reaction. Candidate genes include genes involved in the DNA damage response, programed cell death, inflammation, and angiogenesis. Tumor samples are analyzed by tissue microarrays using immunohistochemistry, denaturing high-performance liquid chromatography, and DNA sequencing to study genetic changes in the tumor.

PROJECTED ACCRUAL: A total of 1,800 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Newly diagnosed or metastatic disease
* Resides within the North Trent Cancer Network (NTCRN) region
* Undergoing therapy at NTCRN centers
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* No concurrent participation in another genetic study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2005-04; Primary Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Correlation of inherited and acquired variations in candidate genes with breast cancer progression and survival

SECONDARY OUTCOMES:
Establishment of a repository of blood and tumor samples

CONTACTS AND LOCATIONS:
Overall Officials: Angela Cox, PhD, Study Chair — University of Sheffield
Locations (1):
- University of Sheffield School of Medicine and Biomedical Sciences, Sheffield, England, United Kingdom